CLINICAL TRIAL: NCT06232499
Title: Effects of Intravenous Laser Irradiation of Blood Treatment With Different Colored Lights on Controlling Recurrent Stroke Risk Factors and Neurological Function in Stroke Patients: a Randomized, Cross-over Trial
Brief Title: Effects of Intravenous Laser Irradiation of Blood Treatment With Different Colored Lights on Controlling Recurrent Stroke Risk Factors and Neurological Function in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Hospital, Ministry of Health and Welfare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 202406
Record Dates: First submitted 2024-01-04; First posted 2024-01-30 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Stroke; Intravenous Laser Irradiation of Blood; Recurrent stroke risk factors
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Red-Blue Arm (Experimental): Participants in this arm first receive 10 sessions of vascular laser treatment with red light, followed by a two-month washout period, and then receive 10 sessions of vascular laser treatment with blue light.
  Interventions: Device: Intravenous Laser Irradiation of Blood
- Blue-Red Arm (Experimental): Participants in this arm first receive 10 sessions of vascular laser treatment with blue light, followed by a two-month washout period, and then receive 10 sessions of vascular laser treatment with red light.
  Interventions: Device: Intravenous Laser Irradiation of Blood

INTERVENTIONS:
Device: Intravenous Laser Irradiation of Blood — The different color lights for Intravenous Laser Irradiation of Blood are red light at 808nm and blue light at 415nm

SUMMARY:
Introduction and Purpose:

Patients with stroke have over a decade of experience with vascular laser treatment. Previous studies predominantly used low-energy vascular lasers with red light, specifically helium-neon lasers with a wavelength of 632.8nm. However, different colored lights are absorbed by cells in the body in varying proportions, leading to potentially different effects. Therefore, there is an interest in understanding the impact of other colored lights on stroke patients. To understand the practical effects of low-energy laser treatment with different colored lights on improving neurological function and controlling recurrent stroke risk factors.

Methods:

A randomized crossover trial will be conducted with a study population consisting of individuals aged 20 and above who have experienced their first stroke within the last 6 months. Exclusion criteria include patients with skin conditions unsuitable for injection or light exposure, those with light allergies, pregnant individuals, those with abnormal blood clotting function, those with implanted pacemakers, and individuals unable to comply with the 5-month study plan. Participants will undergo 10 sessions of infrared light and 10 sessions of blue light vascular laser treatment. Blood tests and neurological assessments will be conducted before each treatment session (10 irradiations) and at the end of the two-month washout period between the two different colored lights. Descriptive analysis and pair t-tests will be employed to compare baseline values between the two groups. Subsequently, repeated measures ANOVA will be used to analyze differences between the intervention group and the control group. The study will examine whether various influencing factors are associated with receiving vascular laser treatment with different colored lights.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as a first-time stroke patient.
2. Onset of illness within 6 months of enrollment.
3. Recruitment period from January to December of the year 113.
4. All participants or their legal representatives must sign the informed consent form.

Exclusion Criteria:

1. Skin diseases that make injection or photosensitivity unsuitable.
2. Pregnancy and abnormal blood clotting function.
3. Presence of a cardiac pacemaker.
4. Inability to comply with the 5-month study plan.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-12-14 (Actual); Study Completion 2024-12-14 (Actual)

PRIMARY OUTCOMES:
Blood urea nitrogen (BUN) test | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  Can reveal whether your urea nitrogen levels are higher than normal, suggesting that your kidneys may not be working properly.
Creatinine test | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  Measure of how well your kidneys are performing their job of filtering waste from your blood.
Uric acid levels | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  Uric acid levels are typically 2.5-7.0 milligrams per deciliter (mg/dL) in males and 1.5-6.0 mg/dL in females. Low levels are rare, but high levels can lead to gout, kidney disease, and other health issues.
Blood cholesterol | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  Indicates blood lipid control
Blood triglycerides | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  Indicates blood lipid control
High-Density Lipoprotein levels | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  Indicates blood lipid control
Low-Density Lipoprotein levels | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  Indicates blood lipid control
Blood Glucose after meal | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  Indicates blood glucose control
Hemoglobin A1c levels | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  Indicates blood glucose control
Complete Blood Count test | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  Indicates blood cell ratio control
Blood Prothrombin Time | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  Indicates blood coagulation function control
Activated Partial Thromboplastin Time levels | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  Indicates blood coagulation function control
Blood Tumor Necrosis Factor-alpha levels | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  Indicates blood Inflammation control
Blood Interleukin-6 levels | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  Indicates blood Inflammation control
High-sensitivity C-reactive Protein levels | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  Indicates blood Inflammation control
Erythrocyte Sedimentation Rate levels | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  Indicates blood Inflammation control
Modified Rankin Scale (MRS) | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  The Modified Rankin Scale is a scale that measures the degree of disability or dependence in daily activities following a neurological event, such as a stroke.
Barthel Index and IADL (Instrumental Activities of Daily Living) Scores | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  Assesses a person's ability to perform basic activities of daily living (ADL), such as bathing, dressing, and feeding. Instrumental Activities of Daily Living extends the assessment to more complex activities, including managing finances and using transportation.
MMSE (Mini-Mental State Examination) Score | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  MMSE is a widely used screening tool for cognitive impairment. It evaluates various cognitive functions, including orientation, memory, and language. Changes in MMSE scores may indicate alterations in cognitive abilities, providing insights into the impact of interventions on cognitive function.
Berg Balance Test Score | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  The Berg Balance Test assesses a person's balance and risk of falling. It includes tasks such as standing on one foot and turning around. Changes in Berg Balance Test scores can indicate improvements or declines in balance and stability.
Fugl-Meyer Assessment Score | before treatment, two weeks after trial began, 2 months and two weeks after trial began, 3 months after trial began, 5 months after trial began
  The Fugl-Meyer Assessment is commonly used to evaluate motor recovery after stroke.
  It assesses motor function, balance, and sensation. Changes in Fugl-Meyer scores can indicate improvements or declines in motor function and overall recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Hospital, Ministry of Health and Welfare, New Taipei City, ROC, Taiwan

IPD SHARING:
Plan to Share IPD: No